CLINICAL TRIAL: NCT04669808
Title: An Open Label, Dose Escalation Study to Evaluate the Safety and Efficacy of Localized Injection of STP705 in Adult Patients With Basal Cell Carcinoma
Brief Title: Open Label, Dose Escalation Study for the Safety and Efficacy of STP705 in Adult Patients With Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-705-006
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Basal Cell Carcinoma
Keywords: BCC; STP705; Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Participants in the first cohort will attend the study center once weekly for an injection of STP705 into the BCC lesion. The participants will receive injections of STP705 once a week for 6 weeks. The clinician will evaluate the change in tumor size at each treatment visit. At the End of Treatment visit, the residual tumor, or former tumor location, will be excised for analysis.
  In the absence of dose limiting toxicities (DLT), the subsequent cohorts will receive increasing doses of STP705, following the same schedule of administration as the first cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A: STP705 30 μg dose (Experimental): Cohort A: STP705 30 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort B: STP705 60 μg dose (Experimental): Cohort B: STP705 60 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort C: STP705 90 μg dose (Experimental): Cohort C: STP705 90 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort D: STP705 120 μg dose (Experimental): Cohort D: STP705 120 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort E: STP705 180 μg dose (Experimental): Cohort E: STP705 180 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort F: STP705 240 μg dose (Experimental): Cohort F: STP705 240 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705
- Cohort G: STP705 320 μg dose (Experimental): Cohort G: STP705 320 μg dose, localized injection, given once a week for 6 weeks
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — Dry powder for intra-and peri-lesional injection.
  Other Names: STP705 Powder for Injection

SUMMARY:
This phase 2, open label, dose escalation study is designed to evaluate the safety, tolerability and efficacy of various doses of STP705 administered as localized injection in patients with Basal Cell Carcinoma (BCC).

Goals:

* To determine the safe and effective recommended dose of STP705 for the treatment of basal cell carcinoma.
* Analysis of biomarkers common to BCC formation pathway including TGF-β1 and COX-2.

DETAILED DESCRIPTION:
Basal cell carcinoma occurs most often on areas of the skin that are exposed to the sun, such as head and neck. The most commonly found clinical feature of Basal Cell Carcinoma (BCC) is an elevated tumor with a pearly and translucent margin and telangiectasia. The color may vary widely from nearly normal skin color to erythematous to violaceous and may also be pigmented. BCC may also resemble noncancerous skin conditions such as eczema or psoriasis. The majority of these cancers occur on areas of skin that are regularly exposed to sunlight or other ultraviolet radiation.

The STP705 drug substance (STP705) is composed of two siRNA oligonucleotides, targeting the expression of TGF-β1 and Cox-2 mRNA respectively. Along with the HKP-enhanced delivery system, the combination is expected to downregulate TGF-β1 and COX-2 expression resulting in the inhibition of tumor growth and provide an alternative non-invasive approach for the treatment of BCC.

This phase 2, open label, dose escalation study is designed to evaluate the safety, tolerability and efficacy of various doses of STP705 administered as localized injection in patients with BCC. This study seeks to establish a safe and effective recommended dose of STP705 for the treatment of BCC. The clinician will evaluate the change in tumor size at each treatment visit. At the End of Treatment visit, the residual tumor, or former tumor location, will be excised for analysis. Expression of biomarkers common to the BCC formation pathway, including TGF-β1 and COX-2, will be evaluated.

Safety and tolerability will be assessed by the number of incidence of adverse events (AEs) and serious adverse events (SAEs); the incidence of AEs and SAEs leading to discontinuation of trial medication; the incidence and severity of Local Skin Response (LSR); hypopigmentation and hyperpigmentation following treatment; and the tolerability of repeated localized administration of STP705 as assessed by investigator-evaluation of injection site reactions for all patients and within each cohort.

The study plans to enroll approximately 35 adult patients at up to 3 clinical sites in the United States. The 35 patients will be divided equally among 7 cohorts (30, 60, 90, 120, 180, 240, and 320 μg dose level) of 5 patients each.

ELIGIBILITY:
Inclusion Criteria: Subjects are required to meet all of the following criteria for enrollment into the study:

1. Male or female adult ≥ 18 years of age.
2. Primary, histologically confirmed trunk or extremity (non-peri-orbital/-anogenital/-facial/-scalp) basal cell carcinoma lesion suitable for excision with a minimum diameter of 0.5 cm and with a maximum diameter of 2.0 cm.
3. Histological diagnosis made no more than 6 months prior to the screening visit.
4. Histological biopsy removed ≤25% of the original volume of the target lesion.
5. No other dermatological disease in the BCC target site or surrounding area, which in the opinion of the investigator, could interfere with the study.
6. Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period.
7. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study.
8. Laboratory values for the tests (listed in the Study Schedule) within the reference ranges as defined by the central laboratory, or "out of range" test results that is clinically acceptable to the investigator. Ability to follow study instructions and likely to complete all study requirements.
9. Written informed consent obtained, including consent for tissue to be examined and stored by the Central Histology Lab.
10. Written consent to allow photographs of the target BCC lesion to be used as part of the study data and documentation.
11. For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral / implant/ injectable/ transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy).

Exclusion Criteria:

1. Pregnant or lactating.
2. Presence of known or suspected systemic cancer.
3. Histological evidence of SCC, or any other non-BCC tumor in the biopsy specimen.
4. Histological evidence of infiltrative or other aggressive histological subtype growth patterns in the biopsy specimen.
5. History of recurrence of the target BCC lesion.
6. Evidence of dermatological disease or confounding skin condition with in 2 cm margin of the target BCC lesion, e.g., SCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa.
7. Concurrent disease or treatment that suppresses the immune system;
8. Patients with baseline QTC > 480 msec using Frederica's formula.
9. Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk.
10. Known sensitivity to any of the ingredients in the study medication.
11. Use of a tanning beds or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the study.
12. Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit.
13. Use of systemic retinoids within the 6 months prior to the screening period.
14. Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period.
15. Use of topical immunomodulators within 2 cm of the target BCC lesion within the 4 weeks prior to the screening period.
16. Treatment with the following topical agents within 2 cm of the target BCC lesion within the 4 weeks prior to the screening visit: amino-levulinic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, ingenol mebutate, or imiquimod.
17. Treatment with liquid nitrogen, surgical excision (excluding diagnostic incisional biopsy) or curettage within 2 cm of the target BCC lesion during the 4 weeks prior to the screening visit.
18. Evidence of current chronic alcohol or drug abuse.
19. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit.
20. In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.
21. Taking any other investigational product within 1 month of first dose of STP705.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with histological clearance of treated basal cell carcinoma lesion at the End of Treatment (EOT) | 6 weeks
  Histological clearance (HC) will be defined as the absence of detectable evidence of BCC tumor cell nests as determined by central pathology review.

SECONDARY OUTCOMES:
Change in clinical diameter of the treated basal cell carcinoma lesion over the 6 week treatment period | over the 6 week treatment period
  A base line assessment of lesion clinical diameter will be made by investigator at T1 (first visit). The change in size will be assessed every week until the surgical excision of BCC at the End of Treatment (EOT) visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No